CLINICAL TRIAL: NCT01271608
Title: Intramuscular and Subcutaneous Injections: is it Necessary to Have Needles Exchanged?
Brief Title: Study to Evaluate the Need of Needle Change for Application of Intramuscular, Subcutaneous and Intradermal Injection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital M'Boi Mirim (Other)
Responsible Party: Luiz Carlos Ribeiro Lamblet/ Nurse, Hospital M Boi Mirim
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE-0203.0.028.000-08
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2009-06

CONDITIONS: Knowledge, Attitudes, Practice; Injection Site Reactions
Keywords: Accident prevention; Blood-borne pathogens; Protective devices.; Needlestick injuries; Injections subcutaneous; Injections intradermal
MeSH Terms: conditions — Behavior; Injection Site Reaction; Needlestick Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: needle exchange — Comparing the pain intensity on a numeric scale (0-10) with intramuscular and subcutaneous injection between a retractable fixed syringe needle and the technique involving needle exchange; Comparing bruise formation following administration of insulin subcutaneous injections between retractable fixed needle and the conventional technique.

SUMMARY:
Comparing the pain intensity on a numeric scale (0-10) with intramuscular and subcutaneous injection between a retractable fixed syringe needle and the technique involving needle exchange; Comparing bruise formation following administration of insulin subcutaneous injections between RFS and the conventional technique.

Method Study site A clinical trial was conducted in two medical-surgical units in a hospital in the period from June 15th to November 30th, 2009, after approval by the Ethics and Research Committee.

Intervention In a group of patients the investigators used syringes with retractable fixed needle to administer subcutaneous and intramuscular injections. In the group of control, the investigators used the standard technique to administer medications.

Population of study Patients were sequentially enrolled through a lottery system of exposure using random numbers kept in sealed, opaque envelopes.

Sampling design and sample size Subcutaneous injection The sample size was based on the expected proportion of bruising following the injection. It was expected that 40% of patients would show bruising with the conventional technique and 20% with the technique under study for subcutaneous applications. With an alpha error of 5% (p = 0.05) and power of study of 80% (beta error of 20% or 0.2) 240 patients were included, 120 in each group.

Intramuscular injection The sample size was based on the proportion of patients with moderate to severe pain. It was considered normal the incidence of moderate to severe pain in 30% with a needle exchange, whereas it was considered an increase of up to 40% with the retractable fixed needle. The investigators included 500 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* The investigators included all patients over 18 who agreed to participate in the study for subcutaneous and intramuscular injections. The monitoring was done after the reading, comprehension check, and signing of the Term of Free Consent and Clarification.

Exclusion Criteria:

* The investigators excluded patients taking anticoagulants or those who had coagulation disorders, injuries, or skin changes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos R Lamblet, Nurse, Principal Investigator — Conselho Regional de Enfermagem de São Paulo
Locations (1):
- M Boi Mirim Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lamblet LC, Meira ES, Torres S, Ferreira BC, Martucchi SD. Randomized clinical trial to assess pain and bruising in medicines administered by means of subcutaneous and intramuscular needle injection: is it necessary to have needles changed? Rev Lat Am Enfermagem. 2011 Sep-Oct;19(5):1063-71. doi: 10.1590/s0104-11692011000500002. English, Portuguese, Spanish. PMID 22030569